CLINICAL TRIAL: NCT04927195
Title: A Ph1a/1b, First in Human, Participant and Investigator-blind Sponsor-unblinded Randomized Placebo-controlled Multiple Dose Study of EDP1867 in Healthy Volunteers & Participants With Moderate Atopic Dermatitis & Optionally, Moderate Psoriasis, and/or Mild Asthma
Brief Title: Study in Healthy Participants and Participants With Moderate Atopic Dermatitis & Optionally, Moderate Psoriasis, and/or Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evelo Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDP1867-101
Record Dates: First submitted 2021-04-15; First posted 2021-06-15 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-03

CONDITIONS: Atopic Dermatitis; Psoriasis; Asthma
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis; Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 12 healthy volunteers; 8 on EDP1867, 4 on placebo. Dose = upto 7.5 x 10^11 cells, capsules, once daily, 14 days total
  Interventions: Drug: EDP1867; Drug: Placebo
- Cohort 2 (Experimental): 12 healthy volunteers; 8 on EDP1867, 4 on placebo. Dose = upto 1.5 x 10^12 cells, capsules, once daily, 14 days total
  Interventions: Drug: EDP1867; Drug: Placebo
- Cohort 3 (Experimental): 24 subjects with moderate atopic dermatitis; 16 on EDP1867, 8 on placebo. Dose = 7.5 x 10^11 cells, capsules, once daily, 56 days
  Interventions: Drug: EDP1867; Drug: Placebo
- Cohort 4 (Experimental): 24 subjects with moderate psoriasis; 16 on EDP1867, 8 on placebo. Dose = 7.5 x 10^11 cells, capsules, once daily, 56 days
  Interventions: Drug: EDP1867; Drug: Placebo
- Cohort 5 (Experimental): 24 subjects with mild asthma; 16 on EDP1867, 8 on placebo. Dose = 7.5 x 10^11 cells, capsules, once daily, 56 days
  Interventions: Drug: EDP1867; Drug: Placebo

INTERVENTIONS:
Drug: EDP1867 — EDP1867 is an orally administered, pharmaceutical preparation of a single strain of bacteria
Drug: Placebo — Placebo oral capsule

SUMMARY:
This Phase 1 study will investigate the safety and tolerability of EDP1867 in healthy volunteers, participants with atopic dermatitis, and, optionally, in participants with psoriasis and/or asthma.

DETAILED DESCRIPTION:
This is a phase 1a/1b, first in human, participant and investigator-blind sponsor-unblinded randomized placebo-controlled multiple dose study of EDP1867 in healthy volunteers and participants with moderate atopic dermatitis and, optionally, moderate psoriasis, and/or mild asthma. This study has been designed to investigate the clinical safety and tolerability of EDP1867 in healthy volunteers, participants with atopic dermatitis, and, optionally, in participants with psoriasis and/or asthma.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥ 18 years to 65 years.
2. Participant has a body mass index of ≥ 18 kg/m2 to ≤ 35 kg/m2.
3. Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG monitoring at Screening and at Baseline.

   Additional Inclusion Criteria for Participants with Moderate Atopic Dermatitis
4. Participant has moderate atopic dermatitis with a minimum of 5% and a maximum of 40% BSA involvement, and an IGA score of 2 or 3.
5. Participant has had a confirmed diagnosis of atopic dermatitis for at least 6 months.
6. All participants must be using an emollient and should continue to use this once daily (or more, as needed) for at least 14 days prior to randomisation, and must continue this treatment once daily (or more, as needed) throughout the study.

   Additional Inclusion Criteria for Participants with Moderate Psoriasis
7. Participant has moderate plaque psoriasis with plaque covering BSA of ≥3% and ≤10% and meets both of the following additional criteria:

   1. PASI score of ≥6 and ≤15, and
   2. PGA score of 2 or 3.
8. Participant has a confirmed diagnosis of plaque psoriasis for at least 6 months.

   Additional Inclusion Criteria for Participants with Mild Asthma
9. Participant has a diagnosis of stable asthma for at least six months
10. FeNO of ≥40ppb.
11. FEV1 ≥70% of predicted normal.

Key Exclusion Criteria:

1. Participant has received live attenuated vaccination within 6 weeks prior to Screening or intends to have such a vaccination during the course of the study (non-live vaccines are permitted).
2. Participant requires treatment with an anti-inflammatory drug during the study period.
3. Participant has an active infection (e.g. sepsis, pneumonia, abscess) or has had an infection requiring antibiotic treatment within 6 weeks prior to study intervention administration.
4. Participant has renal or liver impairment
5. Participant has active neoplastic disease or history of neoplastic disease within 5 years of Screening
6. Participant has undergone major surgery within 4 weeks prior to Screening.
7. Any known cardiac abnormality
8. Participant has a known history of human immunodeficiency virus (HIV)
9. Known, active hepatitis A, hepatitis B (HBV), or hepatitis C (HCV) infection
10. Participant with any type of GI tract disease
11. Participants with a history of any serious psychiatric condition; or on therapy for any psychiatric condition
12. The participant has taken any over-the-counter (OTC) or prescription medication, within 14 days prior to baseline (Day -1); or anticipates an inability to abstain from these products for the duration of the study period
13. The participant has a significant history of drug abuse or regular use of illicit drugs or a history of alcohol abuse within 1 year prior to Screening or has tested positive for drugs of abuse or alcohol at Screening or at baseline.
14. The participant has had an acute, clinically significant illness within 30 days prior to the first dose of study intervention.

    Additional Exclusion Criteria for Participants with Atopic Dermatitis
15. Participant is receiving systemic immunosuppressive or non-biologic atopic dermatitis therapy or has received such therapy within 4 weeks prior to Screening.
16. Participant has received treatment with biologic agents within 12 months prior to first dose.
17. Participant continues to use topical medications, other than emollients, that could affect atopic dermatitis 2 weeks prior to the start of dosing.
18. Participant intends to continue to use sunbeds and/or increase their sun exposure significantly from their normal lifestyle

    Additional Exclusion Criteria for Participants with Psoriasis
19. Psoriasis restricted to scalp, palm, and/or soles only.
20. Non-plaque type of psoriasis
21. Participant is receiving systemic immunosuppressive or nonbiologic psoriasis therapy or has received such therapy within 4 weeks prior to Screening
22. Participant has received treatment with biologic agents within 12 months prior to first dose.
23. Participant continues to use topical medications that could affect psoriasis within 2 weeks prior to the start of dosing
24. Participant intends to continue to use sunbeds and/or increase their sun exposure significantly from their normal lifestyle

    Additional Exclusion Criteria for Participants with Asthma
25. History of life-threatening asthma, or a visit to the emergency department for asthma in the 6 months prior to screening, or exacerbation requiring oral corticosteroids within the previous 3 months.
26. Smoker or nicotine user within the 3 months prior to screening; or a previous smoker with a greater than 10 pack year history.
27. Other significant non-reversible pulmonary disease
28. Use of the following medicines within the specified time-frame prior to screening:

    1. Long-acting inhaled β2-agonists: 8 weeks. Note: short-acting inhaled β2-agonists are permitted as required.
    2. Anti-IgE therapy: 6 months
    3. Inhaled corticosteroids: 8 weeks
    4. Oral or Injected corticosteroids: 8 weeks
    5. Intranasal or topical steroids: 4 weeks
    6. Leukotriene antagonists: 2 weeks
    7. Long-acting muscarinic antagonist: 8 weeks
    8. Xanthines (excluding caffeine), anticholinergics, cromoglycates: 1 week.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measured through Adverse Events (AEs) | Day 1 to Day 70
  Number of participants with AEs by seriousness and relationship to treatment
Safety and tolerability measured through lab measurements | Day 1 to Day 70
  Number of participants with clinically significant change from baseline (Day 0) in laboratory values
Safety and tolerability measured through ECG | Day 1 to Day 70
  Number of participants with clinically relevant changes from baseline (Day 0) ECG parameters
Safety and tolerability measured through physical examination | Day 1 to Day 70
  Physical examination will include, at a minimum, assessments of the cardiovascular, respiratory, oral cavity, GI and neurological systems. Height and weight will also be measured and recorded. Number of participants with clinically relevant changes from baseline (Day 0) physical examination parameters
Safety and tolerability measured through vital signs | Day 1 to Day 70
  Blood pressure, pulse rate, respiratory rate, oxygen saturations and temperature will be assessed. Number of participants with clinically relevant changes in vital signs from baseline (Day 0)

SECONDARY OUTCOMES:
Change in EASI score | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the change from baseline in EASI (Eczema Area and Severity Index) score
Percentage change in EASI score | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the percentage change from baseline in EASI (Eczema Area and Severity Index) score
Change in SCORAD score | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the change from baseline in SCORAD (SCORing Atopic Dermatitis) score
Percentage change in SCORAD score | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the percentage change from baseline in SCORAD (SCORing Atopic Dermatitis) score
Change in BSA | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the change from baseline in BSA (Body Surface Area)
Percentage change in BSA | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the percentage change from baseline in BSA (Body Surface Area)
Change in IGA x BSA | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the change from baseline in IGA x BSA [IGA = Investigator's Global Assessment, BSA = Body Surface Area]
Percentage change in IGA x BSA | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the percentage change from baseline in IGA x BSA [IGA = Investigator's Global Assessment, BSA = Body Surface Area]
Change in DLQI score | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the change from baseline in DLQI (Dermatology Life Quality Index) score
Change in POEM score | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the change from baseline in POEM (Patient-Oriented Eczema Measure) score
Change in Pruritis NRS average itch score | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the change from baseline in Pruritis NRS (Numerical Rating Scale) average itch score
Change in Pruritis NRS worst itch score | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using the change from baseline in Pruritis NRS (Numerical Rating Scale) worst itch score
Achievement of EASI-50 | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using achievement of EASI-50 at day 70
Achievement of EASI-75 | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using achievement of EASI-75 at day 70
Achievement of IGA 0 or 1 | Day 1 to Day 70
  The clinical improvement in subjects with atopic dermatitis will be measured using achievement of IGA 0 or 1 at day 70
Change in PASI score | Day 1 to Day 70
  The clinical improvement in subjects with psoriasis will be measured using change from baseline in PASI score (Psoriasis Area and Severity Index Score)
Percentage change in PASI score | Day 1 to Day 70
  The clinical improvement in subjects with psoriasis will be measured using percentage change from baseline in PASI score (Psoriasis Area and Severity Index Score)
Change in LSS | Day 1 to Day 70
  The clinical improvement in subjects with psoriasis will be measured using change from baseline in LSS (Lesion Severity Score)
Change in BSA | Day 1 to Day 70
  The clinical improvement in subjects with psoriasis will be measured using change from baseline in BSA (Body Surface Area)
Percentage change in BSA | Day 1 to Day 70
  The clinical improvement in subjects with psoriasis will be measured using percentage change from baseline in BSA (Body Surface Area)
Change in PGA x BSA | Day 1 to Day 70
  The clinical improvement in subjects with psoriasis will be measured using change from baseline in PGA x BSA [PGA= Physician's Global Assessment; BSA = Body Surface Area)
Percentage change in PGA x BSA | Day 1 to Day 70
  The clinical improvement in subjects with psoriasis will be measured using percentage change from baseline in PGA x BSA [PGA= Physician's Global Assessment; BSA = Body Surface Area)
Change in DLQI | Day 1 to Day 70
  The clinical improvement in subjects with psoriasis will be measured using change from baseline in DLQI (Dermatology Life Quality Index) score
Achievement of PASI-50 | Day 1 to Day 70
  The clinical improvement in subjects with psoriasis will be measured using achievement of PASI-50 at Day 70
Achievement of PASI-75 | Day 1 to Day 70
  The clinical improvement in subjects with psoriasis will be measured using achievement of PASI-75 at Day 70
Achievement of PGA of 0 or 1 | Day 1 to Day 70
  The clinical improvement in subjects with psoriasis will be measured using achievement of PGA of 0 or 1 at Day 70
Change in FeNO | Day 1 to Day 70
  The clinical improvement in subjects with asthma will be measured using change from baseline in FeNO (Fractional exhaled Nitric Oxide)
Percentage change in FeNO | Day 1 to Day 70
  The clinical improvement in subjects with asthma will be measured using percentage change from baseline in FeNO
Change in FEV1 | Day 1 to Day 70
  The clinical improvement in subjects with asthma will be measured using change from baseline in FEV1 (Forced Expiratory Volume)
Percentage change in FEV1 | Day 1 to Day 70
  The clinical improvement in subjects with asthma will be measured using percentage change from baseline in FEV1 (Forced Expiratory Volume)
Change in FVC | Day 1 to Day 70
  The clinical improvement in subjects with asthma will be measured using change from baseline in FVC (Forced Vital Capacity)
Percentage change in FVC | Day 1 to Day 70
  The clinical improvement in subjects with asthma will be measured using percentage change from baseline in FVC (Forced Vital Capacity)
Change in FEV1/FVC ratio | Day 1 to Day 70
  The clinical improvement in subjects with asthma will be measured using change from baseline in FEV1/FVC ratio
Percentage change in FEV1/FVC ratio | Day 1 to Day 70
  The clinical improvement in subjects with asthma will be measured using percentage change from baseline in FEV1/FVC ratio
Change in PEF | Day 1 to Day 70
  The clinical improvement in subjects with asthma will be measured using change from baseline in PEF (Peak Expiratory Flow)
Percentage change in PEF | Day 1 to Day 70
  The clinical improvement in subjects with asthma will be measured using percentage change from baseline in PEF (Peak Expiratory Flow)
Change in number of exacerbations | Day 1 to Day 56
  The clinical improvement in subjects with asthma will be measured using change from baseline in number of exacerbations across the treatment period
Occurrence of any exacerbation | Day 1 to Day 56
  The clinical improvement in subjects with asthma will be measured using the occurrence of any exacerbation during the treatment period
Number of puffs of SABA medication | Day 1 to Day 56
  The clinical improvement in subjects with asthma will be measured using the number of puffs of SABA medication used in the 7 days prior to Day 28 and Day 56
Use of any SABA medication | Day 1 to Day 56
  The clinical improvement in subjects with asthma will be measured using the occurrence of use of any SABA medication during the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Pui Man Leung, MBChB MRCP FFPM DPM, Principal Investigator — MAC Clinical Research
Locations (7):
- United Kingdom (7):
  - MAC Clinical Research Manchester, Manchester, Greater Manchester
  - Medicines Evaluation Unit (MEU), Manchester, Greater Manchester
  - MAC Clinical Research, Blackpool, Lancashire
  - MAC Clinical Research, Liverpool, Merseyside
  - MAC Clinical Research, Cannock, South Staffordshire
  - MAC Clinical Research, Stockton-on-Tees, Teeside
  - MAC Clinical Research, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: No